CLINICAL TRIAL: NCT01127204
Title: Randomized Phase 3 Trial to Evaluate Two Simplified Antiretroviral Treatment Strategies in HIV Infected Children, Treated by Antiretroviral Triple Therapy Before One Year of Age, in Virological Success in Africa (Burkina Faso, Côte d'Ivoire, Rwanda)
Brief Title: Evaluation of Simplified Antiretroviral Treatment Strategies in HIV Infected Children Treated by Antiretroviral (ARV) Before One Year of Age
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); Public Research Centre Health, Luxembourg (Other); Ministry of Foreign Affairs, Luxembourg (Unknown); University of Ouagadougou, Burkina Faso (Other); Programme PAC-CI, Site ANRS-MIE de Côte d'Ivoire (Other); Ministry of Health, Rwanda (Other Government); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); University of Bordeaux (Other); Institut de Sante Publique, d'Epidémiologie et de Développement (Unknown); Université Montpellier (Other); University of Paris 5 - Rene Descartes (Other); Queen Fabiola Children's University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 12206 MONOD; IP.2007.33011.002 (Other Grant/Funding Number: EDCTP)
Record Dates: First submitted 2010-05-19; First posted 2010-05-20 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: HIV Infections
Keywords: HIV; Antiretroviral therapy; Infant; Sub Saharian Africa
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- arm 1 (reference strategy) (Active Comparator): AZT-3TC-LPV/r twice a day
  Interventions: Drug: AZT-3TC-LPV/r twice a day
- arm 2 (simplification strategy) (Experimental): ABC-3TC-EFV once a day
  Interventions: Drug: ABC-3TC-EFV once a day

INTERVENTIONS:
Drug: AZT-3TC-LPV/r twice a day — AZT sirup (10mg/ml): 4 mg/kg or 180 mg/m2 twice daily 3TC sirup (10mg/ml): 4 mg/kg twice daily LPV/r sirup (80/20 mg/ml): 12 mg/kg twice daily
  Arms: arm 1 (reference strategy)
Drug: ABC-3TC-EFV once a day — ABC sirup (20mg/ml): 16 mg/kg once daily in the morning 3TC sirup (10mg/ml): 8 mg/kg once daily in the morning EFV sirup (30mg/ml): 25 mg/kg once daily in the morning before food intake
  Arms: arm 2 (simplification strategy)

SUMMARY:
The MONOD trial aim to evaluate the implementation of early antiretroviral treatment strategies in HIV-infected infants and assess the feasibility and efficacy of simplifying the initial proposed regimen after a successful one year treatment. The initial treatment is AZT-3TC-LPV/r twice a day. After one year, the children will be randomized in one of the following : arm 1-reference AZT-3TC-LPV/r twice daily; arm 2-simplified ABC-3TC-EFV once daily.

The perspective of this project is to identify antiretroviral strategies to improve treatment access and adherence for children in sub-saharian Africa.

ELIGIBILITY:
Inclusion Criteria for antiretroviral treatment initiation:

* infant follow-up in one of the trial site
* HIV-1 infection diagnose by RT PCR after 6 weeks of life
* age between 3 and 12 month at the antiretroviral treatment initiation
* naive of antiretrovirals except if received for the prevention of mother to child HIV transmission
* HB>=7 g/dl, neutrophiles>750/mm3, creatinin<3xULN, TGO and TGP<3xULN
* signed informed consent

Exclusion Criteria for antiretroviral treatment initiation:

* HIV-2 infection or HIV-1/HIV-2 co-infection
* Known intolerance to one of the trial treatment
* HB<7 g/dl, neutrophiles<750/mm3, creatinin>3xULN, TGO or TGP>3xULN

Inclusion Criteria for randomisation at 12 months in the simplification phase:

* age 24 months at most
* virological success define as 2 consecutive indetectable HIV RNA measured by RT PCR at least 3 months apart.

Exclusion Criteria for randomisation at 12 months in the simplification phase:

* virological failure after the first 12 months of antiretroviral treatment

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 161 (Actual)
Dates: Start 2011-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Initial therapeutic cohort: Virological success | 12 months
  survival without virological failure (death or loss of follow-up or virologic failure, i.e. HIV-ARN ≥400 copies/mL on one consecutive sample), analysis of resistance profile.
Randomised simplification phase: Virological success | 25 months
  survival without virological failure (death or loss of follow-up or virologic failure (HIV-ARN ≥400 copies/mL ))from M13 to M25.

SECONDARY OUTCOMES:
Virological success | 12 months
  HIV RNA < 400 copies / mL
Immunological response | 12 and 25 months
  CD4+ lymphocyte absolute count and percentage
Antiretroviral and cotrimoxazol pharmacokinetic parameters | 6, 19 and 25 months
  The following parameters will be measured or calculated: maximal and minimal concentration (Cmax, Cmin), half life (t1/2), Aire Under the Curve (AUC), clearance and volume of distribution, for all antiretroviral (according to treatment arm : AZT, 3TC, LPV, ABC, EFV) and cotimoxazol.
Tolerance | 12 and 25 month
  occurence of grade 3 and 4 adverse events related to the trial treatment, particularly occurence of immune reconstitution inflammatory syndrome
Adherence | 12 and 25 months
  measurement at each protocol visit of the three last days treatment intake to be corelated to the antiretroviral concentration and virological success
Resistance to antiretroviral | 12 and 25 months
  Genotyping to analyse resistance mutation when virological failure

CONTACTS AND LOCATIONS:
Overall Officials: Marguerite Timite-Konan, Principal Investigator — Service de pédiatrie - CHU Yopougon - Abidjan, Côte d'Ivoire; Jules Mugabo, Principal Investigator — Center for Infectious Desease Control - Kigali, Rwanda; Nicolas Meda, Principal Investigator — Université de Ouagadougou - Ouagadougou, Burkina Faso
Locations (4):
- Burkina Faso (2):
  - Service de maladies infectieuses - CHU Charles de Gaulle, Ouagadougou
  - Service de pédiatrie - CHU Yalgado Ouedraogo, Ouagadougou
- Côte d’Ivoire (2):
  - CEPREF, Abidjan
  - FSU abobo-Avocatier, Abidjan

REFERENCES:
- [Derived] Pressiat C, Toni TD, Treluyer JM, Yonaba C, Dahourou DL, Malateste K, Seguin-Devaux C, Leroy V, Hirt D; MONOD ANRS Study Group. High nevirapine levels in breast milk and consequences in HIV-infected child when initiated on antiretroviral therapy. AIDS. 2021 Nov 15;35(14):2409-2410. doi: 10.1097/QAD.0000000000003043. No abstract available. PMID 34723858
- [Derived] Desmonde S, Frank SC, Coovadia A, Dahourou DL, Hou T, Abrams EJ, Amorissani-Folquet M, Walensky RP, Strehlau R, Penazzato M, Freedberg KA, Kuhn L, Leroy V, Ciaranello AL. Cost-Effectiveness of Preemptive Switching to Efavirenz-Based Antiretroviral Therapy for Children With Human Immunodeficiency Virus. Open Forum Infect Dis. 2019 Jun 11;6(7):ofz276. doi: 10.1093/ofid/ofz276. eCollection 2019 Jul. PMID 31334298
- [Derived] Pressiat C, Mea-Assande V, Yonaba C, Treluyer JM, Dahourou DL, Amorissani-Folquet M, Blanche S, Eboua F, Ye D, Lui G, Malateste K, Zheng Y, Leroy V, Hirt D; MONOD Study Group. Suboptimal cotrimoxazole prophylactic concentrations in HIV-infected children according to the WHO guidelines. Br J Clin Pharmacol. 2017 Dec;83(12):2729-2740. doi: 10.1111/bcp.13397. Epub 2017 Sep 20. PMID 28800382
- [Derived] Pressiat C, Amorissani-Folquet M, Yonaba C, Treluyer JM, Dahourou DL, Eboua F, Blanche S, Mea-Assande V, Bouazza N, Foissac F, Malateste K, Ouedraogo S, Lui G, Leroy V, Hirt D. Pharmacokinetics of Efavirenz at a High Dose of 25 Milligrams per Kilogram per Day in Children 2 to 3 Years Old. Antimicrob Agents Chemother. 2017 Jun 27;61(7):e00297-17. doi: 10.1128/AAC.00297-17. Print 2017 Jul. PMID 28483965
- [Derived] Amani-Bosse C, Dahourou DL, Malateste K, Amorissani-Folquet M, Coulibaly M, Dattez S, Emieme A, Barry M, Rouzioux C, N'gbeche S, Yonaba C, Timite-Konan M, Mea V, Ouedraogo S, Blanche S, Meda N, Seguin-Devaux C, Leroy V. Virological response and resistances over 12 months among HIV-infected children less than two years receiving first-line lopinavir/ritonavir-based antiretroviral therapy in Cote d'Ivoire and Burkina Faso: the MONOD ANRS 12206 cohort. J Int AIDS Soc. 2017 Apr 25;20(1):21362. doi: 10.7448/IAS.20.01.21362. PMID 28453240
- [Derived] Dahourou DL, Amorissani-Folquet M, Malateste K, Amani-Bosse C, Coulibaly M, Seguin-Devaux C, Toni T, Ouedraogo R, Blanche S, Yonaba C, Eboua F, Lepage P, Avit D, Ouedraogo S, Van de Perre P, N'Gbeche S, Kalmogho A, Salamon R, Meda N, Timite-Konan M, Leroy V; MONOD Study Group. Efavirenz-based simplification after successful early lopinavir-boosted-ritonavir-based therapy in HIV-infected children in Burkina Faso and Cote d'Ivoire: the MONOD ANRS 12206 non-inferiority randomised trial. BMC Med. 2017 Apr 24;15(1):85. doi: 10.1186/s12916-017-0842-4. PMID 28434406
- [Derived] Dahourou DL, Amorissani-Folquet M, Coulibaly M, Avit-Edi D, Meda N, Timite-Konan M, Arendt V, Ye D, Amani-Bosse C, Salamon R, Lepage P, Leroy V; Monod Anrs 12206 Study Group. Missed opportunities of inclusion in a cohort of HIV-infected children to initiate antiretroviral treatment before the age of two in West Africa, 2011 to 2013. J Int AIDS Soc. 2016 Mar 23;19(1):20601. doi: 10.7448/IAS.19.1.20601. eCollection 2016. PMID 27015798